CLINICAL TRIAL: NCT06901661
Title: Telerehabilitation for Hip and Knee Osteoarthritis. A Randomized Controlled Trial
Brief Title: Telerehabilitation for Hip and Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-IJRB-N202412017
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Telerehabilitation; Osteoarthritis; Randomized controlled trial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis | interventions — Telerehabilitation; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation (Experimental): Receive a remote exercise program for 40 minutes once a week for 5 weeks
  Interventions: Behavioral: Telerehabilitation
- Standard care (Placebo Comparator): Receive a patient education session once a week for 5 weeks
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Telerehabilitation — Exercise program include Warm-up, Targeted muscle Strengthening, Joint mobilization, and Proprioception
  Arms: Telerehabilitation
Behavioral: Standard care — Education session on their pain, disability, and functional activities
  Arms: Standard care

SUMMARY:
Digital health utilization in the form of telerehabilitation is a popular technology that is very little researched for musculoskeletal disorders particularly hip and knee osteoarthritis (OA). The progression of OA will lead to total hip or knee replacement surgery. As a consequence, the advancing aging population leads to an increased burden on the healthcare system due to rising osteoarthritis. That's why, we will conduct a randomized controlled trial to explore the effectiveness of telerehabilitation in hip and knee osteoarthritis. This study will recruit OA patients into control and experimental groups. The control group will receive a patient education while the experimental group will undergo remote exercise sessions. Both groups will receive one supervised session a week for 5 weeks. The pre- and post-outcome measures will be recorded for functional status of hip and knee, muscle strength, and range of motions of the lower extremity. This innovative study will evaluate the effectiveness of a telemedicine intervention applied to a clinical population in Taiwan. The use of telerehabilitation interventions aims to reduce treatment and transportation costs, as well as save time for patients with OA. This digital health approach also helps to alleviate the workload of physiotherapists and rehabilitation doctors in clinics. The findings from this study could broaden the scope for using remote digital technology to assist clinical patients in diverse settings, especially those with limited or no hospital access.

DETAILED DESCRIPTION:
Purpose: To conduct a randomized controlled trial to explore the efficacy of telerehabilitation intervention for 5 weeks in a clinical population with hip and knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with hip or knee osteoarthritis within last one year
2. having sub-acute or chronic symptoms of pain and functional disability
3. living in an area served by high-speed Internet services (at least 512 kb/s in upload)
4. living within an hour driving distance from the treating hospital
5. physically fit to provide a written consent to participate in this study

Exclusion Criteria:

1. taking sedatives, autoimmune, or other medication that can interfere with their exercise program
2. any health issues that could affect the tests or the rehabilitation program, including surgery over the recent six months
3. having diagnosed with cognitive disorders
4. having recent surgery or major postoperative complications

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | The outcome measures will be recorded before and after finish all 5 week of the intervention
  A questionnaire

SECONDARY OUTCOMES:
Muscle strength | The outcome measures will be recorded before and after finish all 5 week of the intervention
  Static muscle strength of hip and knee flexors and extensors
Range of motion | The outcome measures will be recorded before and after finish all 5 week of the intervention
  The Range of motions of hip and knee flexion and extension

OTHER OUTCOMES:
Borg rate of perceived exertion (RPE) | Evaluate every week for 5 weeks during each exercise session of the experimental group
  6-20 points rating, a score ≤11 will be considered as "low fatigue" and >11 as "high fatigue
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | The outcome measures will be recorded before and after finish all 5 week of the intervention
  A questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chou Chen, Dr., Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No